CLINICAL TRIAL: NCT02791906
Title: Targeting Central Pulsatile Hemodynamics in Chronic Kidney Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Julio A. Chirinos, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 823665
Record Dates: First submitted 2016-05-26; First posted 2016-06-07 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic Kidney Diseases; Chronic Kidney Insufficiency; Chronic Renal Diseases; Chronic Renal Insufficiency; Kidney Insufficiency, Chronic; Cardiac Failure; Congestive Heart Failure; Heart Decompensation; Heart Failure, Congestive; Myocardial Failure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Failure | interventions — Ascorbic Acid

ARMS (2):
- ISMN Only (Experimental): Patients receive only ISMN
  Interventions: Drug: ISMN
- ISMN AND Vitamin C (Experimental): Patients receive both ISMN and Vitamin C
  Interventions: Drug: ISMN; Dietary Supplement: Vitamin C

INTERVENTIONS:
Drug: ISMN
Dietary Supplement: Vitamin C
  Arms: ISMN AND Vitamin C

SUMMARY:
Heart failure (HF) is an epidemic and is a major burden on the US healthcare system. The most common cardiovascular endpoint is HF. Thus, novel interventions to prevent HF in chronic kidney disease (CKD) are highly desirable. This study will assess: the variability in the response to isosorbide mononitrate (ISMN) therapy; the degree of change in central hemodynamics and cardiac endpoints through analysis of changes in left ventricle (LV) mass, diffuse myocardial fibrosis, and myocardial systolic and diastolic function.

DETAILED DESCRIPTION:
This is a open label, parallel arm, randomized study of ISMN with or without vitamin C to improve exercise capacity and LV remodeling in CKD. Twenty subjects with CKD will be enrolled in this study and three different daily doses of sustained release isosorbide mononitrate (SR-ISMN) will be administered over time accompanied by a random administration of vitamin C in half of the subjects (500 mg three times daily). Before administration of SR-ISMN, baseline assessments will be performed. These include arterial tonometry, Doppler echocardiography, reflection magnitude measurements, a bicycle exercise test, activity monitoring, cardiac MRI, 24-hour blood pressure monitoring, and blood drawing. After these assessments, a dose of 30 mg of SR-ISMN will be administered daily (either with or without vitamin C) for the first week, 60 mg SR-ISMN for the second week, and 120 mg for the third week. After each week, blood pressure and central hemodynamics will be assessed. The third week visit also includes the bicycle exercise study and initiating the long term dose (60 or 120 mg) of SR-ISMN. In the long-term phase, blood pressure and hemodynamics are assessed at 12-weeks post initiation of the study medication(s). After 24 weeks we will perform the final assessment, which includes the same tests performed during the baseline assessment. Enrollment will take place at the Hospital of the University of Pennsylvania and the Penn Presbyterian Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stage 3
* Elevated left ventricular mass index or LV posterior wall thickness >1.4 cm documented in a clinically indicated echocardiographic or MRI examination within the previous 24 months or electrocardiographic LV hypertrophy
* Stable medical therapy as defined by no addition, removal or change in dosage >100% of Angiotensin-converting-enzyme (ACE) inhibitors, angiotensin receptor blockers, beta-blockers, or calcium channel blockers for > 30 days
* Current therapy with an ACE inhibitor, hydralazine or a statin, all of which have been shown to reduce nitrate tolerance

Exclusion Criteria:

* A clinically- indicated stress test demonstrating significant myocardial ischemia within 1 year of enrollment, not followed by coronary revascularization
* Rhythm other than sinus (i.e., atrial fibrillation)
* Non-cardiac condition limiting life expectancy to <1 year
* Current or anticipated future need for long acting organic nitrate therapy
* Severe aortic or mitral valve disease
* Hypertrophic cardiomyopathy
* Known infiltrative or inflammatory myocardial disease (amyloid, sarcoid)
* Pericardial disease
* Primary pulmonary arteriopathy
* History of myocardial infarction, unstable angina, percutaneous transluminal coronary angiography (PTCA) or coronary artery bypass grafting (CABG) within 60 days, or requirement for either PTCA or CABG at the time of consent
* Resting heart rate (HR) >100 bpm
* A reduced LV ejection fraction (EF<50%)
* Known severe liver disease (AST >3x normal, alkaline phosphatase or bilirubin >2x normal)
* Allergy to ISMN
* Current therapy with phosphodiesterase inhibitors, such as sildenafil, vardanafil or tadalafil
* Therapy with rosiglitazone
* Current pregnancy or a positive urine pregnancy test; women who become pregnant during the study will be discontinued from the trial
* Therapy with warfarin
* History of kidney stones
* History of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Systolic blood pressure <110 mmHg or diastolic blood pressure <40 mmHg;
* Contraindications to a cardiac MRI: (a) Central nervous system aneurysm clips; (b) Implanted neural stimulators; (c) Implanted cardiac pacemaker or defibrillator; (d) Cochlear implant; (e) Ocular foreign body (e.g. metal shavings); (f) Other implanted medical devices: (e.g. drug infusion ports); (g) Insulin pump; (h) Metal shrapnel or bullet; (i) Claustrophobia; (j) Extreme obesity rendering the patient unable to fit into narrow-bore scanners; (k) Unwillingness of the patient to undergo a cardiac MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Chirinos, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening was performed from electronic medical records searcesh for potential study participants, followed by manual review.
Pre-assignment Details: After assessing subjects for eligibility via electronic health record reviews (n=529), 522 were excluded due to not meeting inclusion/exclusion criteria (n=506), not being interested in participating upon telephone interview (n=3) and various other reasons (inability to contact, inability to exercise, scheduling difficulties; n=13).
Groups:
- ISMN Only: Patients receive only ISMN
  ISMN
- ISMN AND Vitamin C: Patients receive both ISMN and Vitamin C
  ISMN
  Vitamin C
Period: Overall Study
Arm/Group | ISMN Only | ISMN AND Vitamin C
Started | 4 | 3
Completed | 2 | 2
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISMN Only | ISMN AND Vitamin C | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.75 (10.65) | 64 (4.36) | 64.43 (7.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in LV Mass
Description: Variability seen in change in LV mass with ISMN administration measured with steady-state free precession cardiac MRI, outcomes reflect the change, in grams
Time Frame: Measured at Baseline Visit and 24 Week Visit
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | ISMN Only | ISMN AND Vitamin C
Number analyzed (Participants) | 2 | 2
grams | 24.95 (31.5) | -10.4 (1.26)

2. Secondary Outcome: Changes in Diffuse Myocardial Fibrosis
Description: Myocardial ECV was assessed using a modified Look-Locker inversion recovery sequence to assess T1 times before and following the IV administration of gadolinium contrast in a mid-ventricular short-axis slice. Parameters for modified Look-Locker inversion recovery were: field of view=340mm2; matrix size=144×192; slice thickness=6mm; repetition time=2.4ms; echo time=1.18ms; flip angle=30 degrees, bandwidth=1000 Hz/pixel, integrated parallel acquisition techniques=2. Myocardial T1measurements were performed before and at several time points (5, 10, 15, and 20-40 min) post-gadolinium administration. Modified Look-Locker inversion recovery was performed with a 5-3-3 schema with (2 inversions, 5 echo times after inversion 1, 3 T1 recovery heartbeats, and 3 echo times after inversion 2). All T1 measurements were used to compute lambda (the myocardium-blood partition coefficient) as the slope of the myocardial 1/T1 over the blood 1/T1 change, by linear regression.
Time Frame: Measured at Baseline Visit and 24 Week Visit
Population: Patients who had measurements at baseline and 24 weeks.
Measure: Mean (Standard Deviation); unit: % of myocardial tissue composed of ECV
Arm/Group | ISMN Only | ISMN AND Vitamin C
Number analyzed (Participants) | 2 | 2
% of myocardial tissue composed of ECV | -0.68 (4.56) | 2.12 (2.99)

3. Secondary Outcome: Changes in Myocardial Systolic and Diastolic Function
Description: Variability in changes in myocardial function with ISMN administration, assessed via systolic longitudinal strain (measured with tissue tracking MRI) with adequate data for tissue tracking. Strain is the shortening during contraction, expressed as a promotion of the end-diastolic myocardial length. Shortening is indicated by a negative value. Strain is a unit-less metric and is thus expressed in %. A change with negative sign indicates more pronounced shortening of baseline compared to 6 months; a change with positive sign indicates less pronounced shortening during contraction.
Time Frame: Measured at Baseline Visit and 24 visits
Population: patients who underwent measurements at baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: Percent shortening
Arm/Group | ISMN Only | ISMN AND Vitamin C
Number analyzed (Participants) | 2 | 1
Percent shortening | -3.95 (9.67) | 7.23 (0)

4. Secondary Outcome: Pulse Wave Reflection Magnitude
Description: Measured by arterial tonometry and echocardiography. The data reflects estimated changes in each group utilizing all available measurements, collected at all timepoints (baseline visit and weeks 1, 2, 3, 12, and 24 visits). Numbers are estimated changes in each group utilizing available measurements. The change represents the absolute change in the ratio of backward to forward wave amplitudes, multiplied by 100.
Time Frame: Measured between Baseline Visit-Week 24
Population: participants with measurements available at baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % of change in magnitude
Arm/Group | ISMN Only | ISMN AND Vitamin C
Number analyzed (Participants) | 2 | 2
% of change in magnitude | 0.47 (6.11) | -2.28 (8.77)

5. Secondary Outcome: Aerobic Capacity
Description: Variability in changes in aerobic capacity (peak oxygen consumption during maximal supine bicycle exercise test)
Time Frame: Change from Baseline at Week 24 reported
Population: Only 3 subjects had sufficient data to compute a change from baseline, 1 in the ISMN only arm and 2 in the ISMN + Vit C arm. Below are the results of the data that was analyzed for those subjects.
Measure: Mean (Standard Deviation); unit: L of O2 consumed/ minute
Groups:
- ISMN Only: Monotherapy with isosorbide mononitrate
- ISMN AND Vitamin C: Combination therapy with isosorbide mononitrate and vitamin C
Arm/Group | ISMN Only | ISMN AND Vitamin C
Number analyzed (Participants) | 1 | 2
L of O2 consumed/ minute | 0.05732 (0) | 0.32813 (0.49521)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ISMN Only | ISMN AND Vitamin C
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISMN Only (N=4) | ISMN AND Vitamin C (N=3)
Urosepsis requiring hospitalization (Infections and infestations) | 0 (0) | 1 (1) — Participant presented with with bilateral flank pain and chills, acute kidney injury, leukocytosis and E. coli bacteremia. The diagnosis was urosepsis, which was successfully treated with antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISMN Only (N=4) | ISMN AND Vitamin C (N=3)
Worsening renal AKI + Hyperkalemia (Renal and urinary disorders) | 1 (1) | 0 (0)
2n degree AV block (Cardiac disorders) | 0 (0) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Hypokalemia (Renal and urinary disorders) | 1 (1) | 0
fatigue (General disorders) | 0 (0) | 1 (1)
Drowsiness/dizziness/lightheadedness (Nervous system disorders) | 2 (3) | 1 (1)
dry mouth (General disorders) | 1 (1) | 1 (1)
Ankle swelling (Cardiac disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 2 (2)
Headache (General disorders) | 0 (0) | 2 (3)
Balance problems (General disorders) | 0 (0) | 1 (1)
Heart burn (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sleep (General disorders) | 0 (0) | 1 (1)
Sweating (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT02791906/Prot_SAP_000.pdf